CLINICAL TRIAL: NCT07332845
Title: Symmetrical Scapula-pelvis Proprioceptive Neuromuscular Facilitation and Superficial Back Line in Chronic Neck Pain With Hamstring Tightness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Karachi (Other)
Collaborators: Sindh Institute of Physical Medicine and Rehabilitation (Other)
Responsible Party: Principal Investigator, Aftab Ahmed Mirza Baig,DPT, MSAPT, Principal Investigator, University of Karachi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IBC KU-544/2025
Record Dates: First submitted 2025-12-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Chronic Neck Pain; Hamstring Muscle Tightness; Neck Pain
Keywords: neck ache; Exercise; Muscle Stretching; Muscle Inhibition; PNF
MeSH Terms: conditions — Neck Pain; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Data analyst was also blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Symmetrical Scapula-Pelvis Pattern Exercises (Experimental): This arm will receive PNF Dynamic Reversal of Antagonists using Symmetrical Scapula-Pelvis Patterns
  Interventions: Other: Symmetrical Scapula-Pelvis Patterns Exercises
- Control Treatment (Active Comparator): This arm will receive evidence based treatment, the suboccipital muscle inhibition with static stretching of the hamstrings.
  Interventions: Other: Suboccipital muscle inhibition technique; Other: Static stretching of hamstring muscle

INTERVENTIONS:
Other: Suboccipital muscle inhibition technique — The Suboccipital Muscle Inhibition technique is a manual therapy method used by practitioners to relieve tension in the suboccipital muscles, which are located at the base of the skull.
  Arms: Control Treatment
Other: Symmetrical Scapula-Pelvis Patterns Exercises — Symmetrical scapula-pelvis patterns refer to a balanced, aligned posture and movement of the shoulder blades and pelvis which is often a therapeutic goal in physical rehabilitation with proprioceptive neuromuscular facilitation.
  Arms: Symmetrical Scapula-Pelvis Pattern Exercises
Other: Static stretching of hamstring muscle — Static stretching for hamstrings involves holding a position that creates tension in the back of the thigh for 30 seconds.
  Arms: Control Treatment

SUMMARY:
A research study will be conducted at Physiotherapy department of the Sindh Institute of Physical Medicine and Rehabilitation, Karachi, Pakistan. Overall 156 patients with 18-40 years old individuals with neck pain will be eligible and they will be included through non-probability, purposive sampling technique. The written informed consent will be taken from all the patients. They will be divided through Simple random sampling (computer generated software) method into two groups, 78 in each group. Group A (experimental group) will receive PNF Symmetrical Scapula-Pelvis Patterns (PNF-SSPP), group B (control group) will receive sub occipital muscle inhibition technique (SMI) and static stretching (SS) of hamstring muscle. All participants will be assessed using assessment form. Outcome measures will be Pain, disability, disability, neck range of motions, hamstring tightness, head posture, and levator scapulae index. An independent assessor blinded to the treatment will assess all the patients for treatment outcome assessment at baseline, after first session and post treatment. Treatment sessions will be given thrice a week for 6 weeks.

DETAILED DESCRIPTION:
A maximum drop-out rate of 20% is expected. The Statistical package for the social sciences (SPSS) 23 version will be used for data analysing. The Mean ± SD will be calculated for quantitative variables like age. The qualitative variables will be shown through calculated frequencies and percentages. The outcome results of the study (decrease pain intensity, improve disability, improve ROM and improve muscle tightness) taken before, after 1st session and after 18th session will be compared and analyzed. The repeated measure of ANOVA will be used as the statistical test. The p-value of 0.05 will be considered as level of significant.

ELIGIBILITY:
Inclusion Criteria:

* Individual with both male and female gender
* Individuals with chronic neck pain (pain for > 3 month)

Exclusion Criteria:

* Any history related to spinal surgery
* Previous administration of epidural injections
* Neck pain due to specific pathology
* Patients with radiculopathy or myelopathy
* Traumatic spinal cord injury
* Neck pain associated with progressive neurological deficit or loss of strength

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 156 (Estimated)
Dates: Start 2026-01-16 (Actual); Primary Completion 2026-10-26 (Estimated); Study Completion 2026-11-26 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity with visual analogue scale for pain at Day 1 | From enrolment to the end of the first treatment session at Day 1.
  The Visual Analogue Scale is a 10 cm line used to measure pain intensity, where the patient marks a point on the line to indicate their pain level, with 0 representing "no pain" and 10 representing "pain as bad as it could possibly be". A score is obtained by measuring the distance from the "no pain" end to the patient's mark, which can be done in centimeters (0-10) or millimeters (0-100). Higher scores indicate greater pain intensity, and this score helps healthcare providers assess severity, which can be categorized as mild (1-3), moderate (4-6), or severe (7-10)
Change in pain intensity with visual analogue scale for pain at 6 weeks | From enrolment to the end of 18 treatment session at 6 weeks
  The Visual Analogue Scale (VAS) is a 10 cm line used to measure pain intensity, where the patient marks a point on the line to indicate their pain level, with 0 representing "no pain" and 10 representing "pain as bad as it could possibly be". A score is obtained by measuring the distance from the "no pain" end to the patient's mark, which can be done in centimeters (0-10) or millimeters (0-100). Higher scores indicate greater pain intensity, and this score helps healthcare providers assess severity, which can be categorized as mild (1-3), moderate (4-6), or severe (7-10).
Change in range of motion with goniometry at Day 1 | From enrolment to the end of first treatment at Day 1
  Goniometry measures the change in range of motion of a joint in degrees by using a goniometer to calculate the joint's angle. The increase in degrees suggests increase in range of motion and decrease suggests decrease in range of motion.
Change in range of motion with goniometry at 6 weeks | From enrolment to the end of 18 treatment sessions at 6 weeks.
  Goniometry measures the change in range of motion of a joint in degrees by using a goniometer to calculate the joint's angle. The increase in degrees suggests increase in range of motion and decrease suggests decrease in range of motion.
Change in neck disability with Neck Disability Index at day 1 | From enrolment to the end of first treatment session at Day 1.
  A change in the Neck Disability Index score indicates a change in a patient's self-reported neck disability. A higher score means greater disability.The NDI is scored from 0 to 50, or 0% to 100%. A score of 0 indicates no limitation, while a score of 50 represents complete limitation.
Change in neck disability with Neck Disability Index at 6 weeks | From enrolment to the end of 18 treatment sessions at 6 weeks.
  A change in the Neck Disability Index score indicates a change in a patient's self-reported neck disability. A higher score means greater disability.The NDI is scored from 0 to 50, or 0% to 100%. A score of 0 indicates no limitation, while a score of 50 represents complete limitation.
Change in hamstring tightness with Sit and Reach (SR) test at Day 1 | From enrolment to the end of first treatment session at Day 1.
  A low Sit and Reach test score in centimetre indicates tight hamstrings, while a higher score shows better hamstring flexibility. When a person with tight hamstrings performs the Sit and Reach test, the muscles pull the pelvis into a posterior tilt, which limits the ability to reach as far and can cause the lower back to round instead of the spine flexing naturally. As hamstring tightness decreases through stretching, the SR score increases, signifying greater flexibility and improved superficial back line.
Change in hamstring tightness with Sit and Reach (SR) test at 6 weeks | From enrolment to the end of 18 treatment sessions at 6 weeks.
  A low Sit and Reach test score in centimetre indicates tight hamstrings, while a higher score shows better hamstring flexibility. When a person with tight hamstrings performs the Sit and Reach test, the muscles pull the pelvis into a posterior tilt, which limits the ability to reach as far and can cause the lower back to round instead of the spine flexing naturally. As hamstring tightness decreases through stretching, the SR score increases, signifying greater flexibility and improved superficial back line.

SECONDARY OUTCOMES:
Change in head posture with goniometry at Day 1 | From enrolment to the end of first treatment session at Day 1
  Goniometry can measure changes in forward head posture by using a goniometer to calculate the craniovertebral angle. This involves placing the goniometer's base on the C7 spinous process and the moving arm on the tragus of the ear, with a smaller CVA angle indicating a greater degree of forward head posture and vice versa. Changes are tracked by taking repeated measurements over time to see if the CVA increases (improving posture) or decreases (worsening posture).
Change in head posture with goniometry at 6 weeks | From enrolment to the end of 18 treatment sessions at 6 weeks
  Goniometry can measure changes in forward head posture by using a goniometer to calculate the craniovertebral angle. This involves placing the goniometer's base on the C7 spinous process and the moving arm on the tragus of the ear, with a smaller CVA angle indicating a greater degree of forward head posture and vice versa. Changes are tracked by taking repeated measurements over time to see if the CVA increases (improving posture) or decreases (worsening posture).
Change in levator scapulae index with vernier caliper at Day 1 | From enrolment to the end of first treatment session at Day 1
  The levator scapulae index is a measurement technique used to assess the relative length of the levator scapulae muscle. It provides a normalized value by comparing the muscle's length to an individual's total body height, which accounts for variations in size between patients. A vernier caliper is the tool used for this measurement due to its accuracy. A normal levator scapulae index range is greater than or equal to 7.44. Decrease in score suggests decrease in muscle length and increase suggests increase in length.
Change in levator scapulae index with vernier caliper at 6 weeks | Time Frame: From enrolment to the end of 18 treatment sessions at 6 weeks
  The levator scapulae index is a measurement technique used to assess the relative length of the levator scapulae muscle. It provides a normalized value by comparing the muscle's length to an individual's total body height, which accounts for variations in size between patients. A vernier caliper is the tool used for this measurement due to its accuracy. A normal levator scapulae index range is greater than or equal to 7.44. Decrease in score suggests decrease in muscle length and increase suggests increase in length.

CONTACTS AND LOCATIONS:
Overall Officials: Aftab Ahmed Mirza Baig, PhD, Principal Investigator — University of Karach; Basit Ansari, PhD, Study Director — University of Karachi
Locations (1):
- Sindh Institute of Physical Medicine and Rehabilitation, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No